CLINICAL TRIAL: NCT01351831
Title: The Difference Between Rehabilitation With or Without Progressive Strength Training After Fast-track Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: The Difference Between Rehabilitation With or Without Strength Training After Total Knee Replacement
Acronym: TKA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Thomas Linding Jakobsen, Research Physiotherapist, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-3-2010-106
Record Dates: First submitted 2011-04-28; First posted 2011-05-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Arthroplasty, Replacement, Knee; Resistance training; Physical Therapy Modalities; Randomized Controlled Trial
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Rehabilitation; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rehabilitation with strength training (Experimental)
  Interventions: Other: Rehabilitation with strength training
- Rehabilitation without strength training (Active Comparator)
  Interventions: Other: Rehabilitation without strength training

INTERVENTIONS:
Other: Rehabilitation with strength training — The rehabilitation programme lasts 1 hour per session, and is performed twice per week for 7 weeks. The rehabilitation program consists of balance-, mobility- and functional training exercises etc. In addition, the participants perform unilateral (operated leg) knee-extensions and leg presses in 2 sets for each strength training exercise, using relative loads of 12 RM (week 1), 10 RM (weeks 2-5), and 8 RM (week 6-7). All sets are performed to failure.
  Arms: Rehabilitation with strength training
Other: Rehabilitation without strength training — The rehabilitation programme lasts 1 hour per session, and is performed twice per week for 7 weeks. The rehabilitation program consists of the same balance-, mobility- and functional training exercises etc. as used in the other experimental arm.
  Arms: Rehabilitation without strength training

SUMMARY:
Background and purpose:

In the early phase after a total knee replacement (TKA), patients experience a decrease in leg muscle strength with up to about 80%. This considerable loss of muscle strength is related to reduced functional performance at this point in time. As the loss of muscle strength and functional performance is most pronounced early after TKA, rehabilitation including strength training initiated early after TKA seems a logical choice. However, tradition and fear of symptom exacerbation, such as increased knee joint swelling, knee pain and slow recovery of knee joint range of motion, have typically precluded strength training early after TKA.

Hypothesis:

Our hypothesis is that the effect of early rehabilitation including strength training will be greater than rehabilitation without strength training. If the hypothesis is confirmed, strength training early after TKA could be implemented directly into clinical rehabilitation practice.

Participants and methods:

Seventy participants with a unilateral TKA, between the age of 18 to 80 years, who understand and speak Danish, have given informed consent, will be included in this study.The study is a single-blinded randomized controlled study, where the participants receive supervised 1) rehabilitation with or 2) rehabilitation without strength training in 7 weeks. All components of the rehabilitation program (balance-, and mobility training etc.) are the same in both groups except the strength training exercises. Instead of the strength training exercises, the group without strength training spend more time on warm-up exercises, mobility- and balance exercises. The rehabilitation program lasts 1 hour per session, and will be performed twice per week. The participants perform a test battery 4 times from before to 6 months after the TKA. The test battery assesses the participants' walking ability, leg strength, knee pain, knee joint swelling- and range of motion, and self-reported function and quality of life.

Ethical issues:

From a pilot study conducted in the beginning of 2010, the investigators found, that strength training initiated early after TKA seems feasible, and does not increase knee joint swelling and knee pain. None of the financial supporters, or any of the authors, have any potential conflicts of interest with regard to the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a primary unilateral total knee arthroplasty.
* Age between 18 and 80 years.
* Participants must understand and speak Danish.
* Participants undergo surgery at Copenhagen University Hospital, Hvidovre, and live in the counties of Copenhagen, Brøndby or Hvidovre.

Exclusion Criteria:

* Disease/Musculoskeletal disorder, which requires special rehabilitation modality.
* Alcohol and drug abuse.
* Lack of wish to participate or unwillingness to sign an informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the maximal distance (in meters) walked in 6 minutes at 2 months after surgery. | Pre-surgery (baseline) and 2 months after surgery (primary endpoint) .
  The 6-minute walk test (6MWT) measures the maximal distance a participant is able to walk in 6 minutes between 2 cones placed 29 meters apart from each other.
  Further assessments: 1 month and 6 months.

SECONDARY OUTCOMES:
Change from baseline in maximum isometric knee-extension and knee-flexion strength at 2 months after surgery. | Pre-surgery (baseline) and 2 months after surgery (primary endpoint).
  Maximum isometric knee-extension and knee-flexion strength of the operated leg are assessed using a computerized strength chair (Good Strength Chair, Metitur Oy, Jyvasklya, Finland.
  Further assessments: 1 month and 6 months.
Change from baseline in maximum concentric leg press power at 2 months after surgery. | Pre-surgery (baseline) and 2 months after surgery (primary endpoint).
  Maximum concentric leg press power of the operated leg is assessed using a leg extensor power rig (Medical Engineering Unit, University of Nottingham - Medical School, Nottingham, UK).
  Further assessments: 1 month and 6 months.
Change from baseline in knee pain during activity and rest at 2 months after surgery. | Pre-surgery (baseline) and 2 months after surgery (primary endpoint).
  Knee pain during activity, and rest before and after examination, are assessed using a 100-mm mechanical Visual Analogue Scale (VAS).
  Further assessments: 1 month and 6 months.
Change from baseline in knee joint swelling at 2 months after surgery. | Pre-surgery (baseline) and 2 months after surgery (primary endpoint).
  Knee joint swelling of the operated leg is assessed by measuring the knee joint circumference with a tape measure.
  Further assessments: 1 month and 6 months
Change from baseline in knee joint range of motion (ROM) at 2 months after surgery. | Pre-surgery (baseline) and 2 months after surgery (primary endpoint).
  Knee joint ROM of the operated leg is assessed using a large universal goniometer.
  Further assessments: 1 month and 6 months.
Change from baseline in self-reported function at 2 months after surgery. | Pre-surgery (baseline) and 2 months after surgery (primary endpoint).
  The self-reported function is assessed using Knee injury and Osteoarthritis Outcome Score (KOOS).
  Further assessments: 1 month and 6 months.
Change from baseline in self-reported function at 2 months after surgery. | Pre-surgery (baseline) and 2 months after surgery (primary endpoint).
  Self-reported function is assessed using Oxford Knee Score (OKS). Further assessments: 1 month and 6 months.
Change from baseline in self-reported quality of life at 2 month after surgery. | Pre-surgery (baseline) and 2 months after surgery (primary endpoint).
  Self-reported quality of life is assessed using EuroQol questionnaire (EQ-5D). Further assessments: 1 month and 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Centre, Copenhagen University Hospital, Hvidovre, Hvidovre, Denmark

REFERENCES:
- [Derived] Langkilde A, Jakobsen TL, Bandholm TQ, Eugen-Olsen J, Blauenfeldt T, Petersen J, Andersen O. Inflammation and post-operative recovery in patients undergoing total knee arthroplasty-secondary analysis of a randomized controlled trial. Osteoarthritis Cartilage. 2017 Aug;25(8):1265-1273. doi: 10.1016/j.joca.2017.03.008. Epub 2017 Mar 16. PMID 28323139
- [Derived] Jakobsen TL, Kehlet H, Husted H, Petersen J, Bandholm T. Early progressive strength training to enhance recovery after fast-track total knee arthroplasty: a randomized controlled trial. Arthritis Care Res (Hoboken). 2014 Dec;66(12):1856-66. doi: 10.1002/acr.22405. PMID 25074397